CLINICAL TRIAL: NCT03083470
Title: Phase 2 Dose-Rising Study of SOR007 Ointment for Actinic Keratosis
Brief Title: Study of SOR007 Ointment for Actinic Keratosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: DFB Soria, LLC (Industry)
Collaborators: US Biotest, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: SOR007-2017-04
Record Dates: First submitted 2017-03-14; First posted 2017-03-20 (Actual); Results first posted 2019-04-25 (Actual); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Actinic Keratosis
MeSH Terms: conditions — Keratosis, Actinic | interventions — Ointments

STUDY DESIGN:
Intervention Model Description: Phase 2, randomized, dose-rising, double-blind trial. Subjects will enroll in four dose-escalating cohorts of eight subjects each. Each cohort will be randomized to SOR007 or Ointment vehicle in a ratio of 3:1. Safety will be assessed in an ongoing manner and formal safety reviews will be conducted four times for each cohort: at Day 8, Day 15, Day 21, and Day 28 for the last subject enrolled in each cohort. The next dose level cohort will enroll upon a finding of safety and tolerability at the previous cohort's second safety review. Once the last cohort has completed the study, all available data, including safety, pharmacokinetics, and preliminary efficacy will be analyzed. The PK blood samples will be analyzed per cohort when the last subject of each cohort completes Day 28.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- SOR007 0.15% (Experimental): SOR007 Ointment 0.15% applied to the face twice daily for 28 days
  Interventions: Drug: SOR007 (Uncoated Nanoparticulate Paclitaxel) Ointment
- SOR007 0.3% (Experimental): SOR007 Ointment 0.3% applied to the face twice daily for 28 days
  Interventions: Drug: SOR007 (Uncoated Nanoparticulate Paclitaxel) Ointment
- SOR007 1.0% (Experimental): SOR007 Ointment 1.0% applied to the face twice daily for 28 days
  Interventions: Drug: SOR007 (Uncoated Nanoparticulate Paclitaxel) Ointment
- SOR007 (Experimental): SOR007 Ointment 2.0% applied to the face twice daily for 28 days
  Interventions: Drug: SOR007 (Uncoated Nanoparticulate Paclitaxel) Ointment
- Ointment Vehicle (Sham Comparator): SOR007 Ointment vehicle applied to the face twice daily for 28 days
  Interventions: Other: SOR007 Ointment Vehicle

INTERVENTIONS:
Drug: SOR007 (Uncoated Nanoparticulate Paclitaxel) Ointment — SOR007 will be applied topically to a target AK lesion test field twice daily for up to 28 days, or until all lesions resolve. The maximum total amount of SOR007 that will be applied daily will be 1 finger-tip unit (FTU), approximately 0.5g. No more than 25cm2, approximately 0.15% of the total body surface area, will be treated.
  Arms: SOR007; SOR007 0.15%; SOR007 0.3%; SOR007 1.0%
Other: SOR007 Ointment Vehicle — SOR007 ointment vehicle will be applied topically to a target AK lesion test field twice daily for up to 28 days, or until all lesions resolve. The maximum total amount of Ointment vehicle that will be applied daily will be 1 finger-tip unit (FTU), approximately 0.5g. No more than 25cm2, approximately 0.15% of the total body surface area, will be treated.
  Arms: Ointment Vehicle

SUMMARY:
A Phase 2, randomized, double-blind, dose rising study to determine the safety, tolerability, and preliminary efficacy of four concentrations of SOR007 (Uncoated Nanoparticulate Paclitaxel) Ointment (SOR007) compared to SOR007 ointment vehicle applied to actinic keratosis (AK) lesions on the face twice daily for up to 28 days.

DETAILED DESCRIPTION:
In this Phase 2, randomized, double-blind, dose rising trial, subjects with actinic keratosis will receive topical application of SOR007 Ointment (in four concentrations) or SOR007 Ointment vehicle to the face twice daily for up to 28 days. Subjects will be enrolled in four dose-escalating cohorts of eight subjects and randomized to SOR0007 or Ointment vehicle in a ratio of 3:1. Cohorts will be enrolled sequentially starting at the lowest concentration.

Safety will be assessed in an ongoing manner and formal safety reviews will be conducted four times for each cohort: at Day 8, Day 15, Day 21, and Day 28 for the last subject enrolled in each cohort. The next dose level cohort will enroll upon a finding of safety and tolerability at the previous cohort's second (Day 15) safety review.

The safety and tolerability of SOR007 will be demonstrated by local toxicity, adverse events, laboratory assessments and vital signs. Subjects will be observed for reduction in the number of AK lesions to determine preliminary efficacy. Plasma samples will be taken at various time points throughout the study to characterize the pharmacokinetics of SOR007.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.
* Men and women with actinic keratosis.
* Age 45-85.
* Women who have had surgical sterilization or are post-menopausal (absence of menses for at least one year) are eligible. Women of child-bearing potential who are non-pregnant, non-nursing, and willing to avoid pregnancy during the course of the study and during the menstrual cycle following completion of their participation in the study are eligible. (Adequate contraception is defined as regular use of diaphragm with condoms, IUD with condoms, or systemic contraceptives if used for at least three months prior to enrollment in the study.) A negative pregnancy test is required as an entry criteria. Women must continue to use the method of contraceptive for at least 30 days after the last administration of study drug.
* Male subjects must agree to sexual abstinence or use adequate contraception when sexually active in combination with their female partners, if they are of childbearing potential. That means the volunteer must be vasectomized or use a condom and his female partner must either be surgically sterile (hysterectomy or tubal ligation) or agree to use a reliable method of contraception with a failure rate of less than 1% per year when used consistently and correctly such as implants, injectables, combined oral contraceptives, or non-DalKon Shield IUDs. This applies from signing of informed consent form until 90 days after the last study drug administration. Methods of contraception must have been effective for at least 30 days on the day of signing of informed consent. Male volunteers must also refrain from sperm donation from the time of singing informed consent form until 90 days after the last study drug administration.
* Presence of 4-8 AK lesions total in a 25 cm2 area identified on the face through transparency mapping and photographs. The face area will be defined from hair line to jaw line. The scalp will not be included. An imaginary normal hair line will be the upper boundary for bald men.
* Able to refrain from the use of all other topical medications to the facial area during the treatment period.
* Considered reliable and capable of understanding their responsibility and role in the study.

Exclusion Criteria:

* History of allergy or hypersensitivity to paclitaxel.
* Lesions that are thicker than 1 mm or larger than 9 mm will not be included in the lesion counts.
* Lesions suspicious for squamous cell carcinoma, basal cell carcinoma, or melanoma will not be included in lesion counts and cannot be in the 25 cm2 area of treatment.
* Abnormal pre-existing dermatologic conditions which might affect the normal course of the disease (e.g. albinism or chronic vesiculobullous disorders).
* Positive urine pregnancy test in women of child-bearing potential.
* Inability to use adequate birth control measures for men or women of child-bearing potential, as defined above.
* Serious psychological illness.
* Significant history within the past year of alcohol or drug abuse.
* During the 30 day period preceding study entry: Participating in any clinical research; using topical paclitaxel for AK; using any other topical agents including but not limited to actinex, glycolic acid products, alpha-hydroxy acid products, and chemical peeling agents for the treatment of AK; using any systemic steroids or topical corticosteroids, having cryosurgery.
* Use of sun lamps or sun tanning beds or booths during the 2 weeks prior to first application and until final visit.
* Prior treatment with systemic paclitaxel or systemic cancer therapy within 6 months of study entry.
* Medical history which, based on the clinical judgment of the Investigator implied an unlikelihood of successful completion of the study.

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2017-05-18 (Actual); Primary Completion 2018-03-12 (Actual); Study Completion 2018-03-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leanne Drummond, Study Director — US Biotest
Locations (1):
- Moore Clinical Research, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- SOR007 0.15%: SOR007 Ointment 0.15% was applied topically to a target AK lesion test field twice daily for up to 28 days, or until all lesions resolved. The maximum total amount of SOR007 applied daily was 1 finger-tip unit (FTU), approximately 0.5g. No more than 25cm2, approximately 0.15% of the total body surface area, was treated.
- SOR007 0.3%: SOR007 Ointment 0.3% was applied topically to a target AK lesion test field twice daily for up to 28 days, or until all lesions resolved. The maximum total amount of SOR007 applied daily was 1 finger-tip unit (FTU), approximately 0.5g. No more than 25cm2, approximately 0.15% of the total body surface area, was treated.
- SOR007 1.0%: SOR007 Ointment 1.0% was applied topically to a target AK lesion test field twice daily for up to 28 days, or until all lesions resolved. The maximum total amount of SOR007 applied daily was 1 finger-tip unit (FTU), approximately 0.5g. No more than 25cm2, approximately 0.15% of the total body surface area, was treated.
- SOR007 2.0%: SOR007 Ointment 2.0% was applied topically to a target AK lesion test field twice daily for up to 28 days, or until all lesions resolved. The maximum total amount of SOR007 applied daily was 1 finger-tip unit (FTU), approximately 0.5g. No more than 25cm2, approximately 0.15% of the total body surface area, was treated.
- Ointment Vehicle: SOR007 Ointment vehicle was applied topically to a target AK lesion test field twice daily for up to 28 days, or until all lesions resolved. The maximum total amount of SOR007 applied daily was 1 finger-tip unit (FTU), approximately 0.5g. No more than 25cm2, approximately 0.15% of the total body surface area, was treated.
Period: Overall Study
Arm/Group | SOR007 0.15% | SOR007 0.3% | SOR007 1.0% | SOR007 2.0% | Ointment Vehicle
Started | 6 | 6 | 6 | 6 | 9
Completed | 6 | 6 | 6 | 6 | 7
Not Completed | 0 | 0 | 0 | 0 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SOR007 0.15% | SOR007 0.3% | SOR007 1.0% | SOR007 2.0% | Ointment Vehicle | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 9 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.2 (6.24) | 67.5 (8.07) | 62.3 (7.31) | 62.2 (11.84) | 62.6 (7.65) | 64.4 (8.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 4 | 5 | 6 | 20
  Male | 2 | 5 | 2 | 1 | 3 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 2 | 0 | 2 | 4
  Not Hispanic or Latino | 6 | 6 | 4 | 6 | 7 | 29
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 6 | 6 | 6 | 6 | 9 | 33
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 6 | 6 | 9 | 33

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events
Description: Treatment emergent adverse events including all reported adverse events, laboratory assessments, physical examination findings, and vital signs.
Time Frame: 56 days
Measure: Count of Participants; unit: Participants
Arm/Group | SOR007 0.15% | SOR007 0.3% | SOR007 1.0% | SOR007 2.0% | Ointment Vehicle
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 9
Participants | 2 | 1 | 3 | 1 | 1

2. Secondary Outcome: Pharmacokinetics: Area Under the Plasma Concentration Versus Time Curve (AUC) of SOR007
Description: Pharmacokinetic (PK) samples were taken on Day 1 at 1h, 2h, 4h, and 6h post application; on Day 8, Day 15, and Day 21 after the first daily application; and on Day 28 at 1h, 2h, 4h, 6h, and 12h after the first daily application.
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: pg·hr/mL
Arm/Group | SOR007 0.15% | SOR007 0.3% | SOR007 1.0% | SOR007 2.0% | Ointment Vehicle
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 9
pg·hr/mL | NA (NA) — Plasma paclitaxel concentrations were generally near the limit of quantitation (10 pg/mL). Paclitaxel pharmacokinetic parameters could only be determined on Day 28 in three of the six patients treated with 2% SOR007 Ointment. | NA (NA) — Plasma paclitaxel concentrations were generally near the limit of quantitation (10 pg/mL). Paclitaxel pharmacokinetic parameters could only be determined on Day 28 in three of the six patients treated with 2% SOR007 Ointment. | NA (NA) — Plasma paclitaxel concentrations were generally near the limit of quantitation (10 pg/mL). Paclitaxel pharmacokinetic parameters could only be determined on Day 28 in three of the six patients treated with 2% SOR007 Ointment. | 180 (45.0) | NA (NA) — Plasma paclitaxel concentrations were generally near the limit of quantitation (10 pg/mL). Paclitaxel pharmacokinetic parameters could only be determined on Day 28 in three of the six patients treated with 2% SOR007 Ointment.

3. Secondary Outcome: Pharmacokinetics: Peak Plasma Concentration (Cmax) of SOR007
Description: as for outcome 2
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | SOR007 0.15% | SOR007 0.3% | SOR007 1.0% | SOR007 2.0% | Ointment Vehicle
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 9
pg/mL | NA (NA) — Plasma paclitaxel concentrations were generally near the limit of quantitation (10 pg/mL). Paclitaxel pharmacokinetic parameters could only be determined on Day 28 in three of the six patients treated with 2% SOR007 Ointment. | NA (NA) — Plasma paclitaxel concentrations were generally near the limit of quantitation (10 pg/mL). Paclitaxel pharmacokinetic parameters could only be determined on Day 28 in three of the six patients treated with 2% SOR007 Ointment. | NA (NA) — Plasma paclitaxel concentrations were generally near the limit of quantitation (10 pg/mL). Paclitaxel pharmacokinetic parameters could only be determined on Day 28 in three of the six patients treated with 2% SOR007 Ointment. | 18.3 (3.61) | NA (NA) — Plasma paclitaxel concentrations were generally near the limit of quantitation (10 pg/mL). Paclitaxel pharmacokinetic parameters could only be determined on Day 28 in three of the six patients treated with 2% SOR007 Ointment.

4. Secondary Outcome: Pharmacokinetics: Time at Which Peak Plasma Concentration is Observed (Tmax) of SOR007
Description: as for outcome 2
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | SOR007 0.15% | SOR007 0.3% | SOR007 1.0% | SOR007 2.0% | Ointment Vehicle
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 9
hr | NA (NA) — Plasma paclitaxel concentrations were generally near the limit of quantitation (10 pg/mL). Paclitaxel pharmacokinetic parameters could only be determined on Day 28 in three of the six patients treated with 2% SOR007 Ointment. | NA (NA) — Plasma paclitaxel concentrations were generally near the limit of quantitation (10 pg/mL). Paclitaxel pharmacokinetic parameters could only be determined on Day 28 in three of the six patients treated with 2% SOR007 Ointment. | NA (NA) — Plasma paclitaxel concentrations were generally near the limit of quantitation (10 pg/mL). Paclitaxel pharmacokinetic parameters could only be determined on Day 28 in three of the six patients treated with 2% SOR007 Ointment. | 1.33 (2.31) | NA (NA) — Plasma paclitaxel concentrations were generally near the limit of quantitation (10 pg/mL). Paclitaxel pharmacokinetic parameters could only be determined on Day 28 in three of the six patients treated with 2% SOR007 Ointment.

5. Secondary Outcome: Percent Change in Number of AK Lesions
Description: AK lesions in the target test field were photographed and tracings were created at baseline and at subsequent visits to track whether lesions were clear or still present.
Time Frame: Baseline and 56 days
Population: Two subjects, both receiving Vehicle, were withdrawn early from the study; one of these subjects participated long enough to be included in the analysis of the efficacy endpoint and one did not. Therefore, there are 8 subjects in the Ointment Vehicle arm of the study.
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | SOR007 0.15% | SOR007 0.3% | SOR007 1.0% | SOR007 2.0% | Ointment Vehicle
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8
Percent Change | -34.68 (27.432) | -34.72 (27.576) | -53.06 (18.868) | -58.33 (30.277) | -48.75 (22.321)

6. Secondary Outcome: Percent Change in Size of AK Lesions
Description: Percent change in size of AK lesions was determined with measurements obtained at Baseline and 56 days. A measurement was also obtained at Day 28, but was not used to calculated percent change for the purposes of this outcome measure.
Time Frame: Baseline and 56 days
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | SOR007 0.15% | SOR007 0.3% | SOR007 1.0% | SOR007 2.0% | Ointment Vehicle
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8
Percent Change | -46.20 (25.698) | -35.83 (17.811) | -58.12 (15.989) | -62.32 (27.544) | -59.22 (24.169)

ADVERSE EVENTS:
Time Frame: 56 Days
Arm/Group | SOR007 0.15% | SOR007 0.3% | SOR007 1.0% | SOR007 2.0% | Ointment Vehicle
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/9
Other Adverse Events (participants affected / at risk) | 2/6 | 1/6 | 3/6 | 1/6 | 1/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | SOR007 0.15% (N=6) | SOR007 0.3% (N=6) | SOR007 1.0% (N=6) | SOR007 2.0% (N=6) | Ointment Vehicle (N=9)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Impaired healing (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Breast Pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0/0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0/0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-04-20): https://cdn.clinicaltrials.gov/large-docs/70/NCT03083470/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-03): https://cdn.clinicaltrials.gov/large-docs/70/NCT03083470/SAP_001.pdf